CLINICAL TRIAL: NCT06034080
Title: DISAPEAR Trial: Interventions to De-implement Unnecessary Antibiotic Prescribing for Children With Ear Infections
Brief Title: Interventions to De-implement Unnecessary Antibiotic Prescribing for Children With Ear Infections
Acronym: DISAPEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: AllianceChicago (Other); Mayo Clinic (Other); Patient-Centered Outcomes Research Institute (Other); Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-1096; IHS-2022C2-28005 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Otitis Media; Ear Infection; Pediatric Infectious Disease
Keywords: Shared Decision-Making; Health-System Level Intervention
MeSH Terms: conditions — Otitis Media; Otitis | interventions — SDM; Educational Status

STUDY DESIGN:
Intervention Model Description: Mutli-Center Cluster Randomized Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health System Level (HSL) Intervention (Active Comparator): The HSL Intervention is based on the CDC Core Elements of Stewardship and the HSL intervention is recommended by national guidelines. Sites randomized to this arm will require:
  1. A change in their Electronic Health Record to their prescription fields to align with national guidelines
  2. Individualized feedback report to their clinicians and clinic overall
  3. And virtual learning sessions and continuing medical education credits for clinicians.
  Interventions: Other: Changes to the electronic health record (EHR); Other: Individualized audit and feedback reporting for clinicians; Other: Clinician education sessions
- Hybrid Intervention (Experimental): The Hybrid Intervention will be comprised of Shared Decision-Making (SDM) and the HSL Intervention. A previously validated SDM aid for ear infection care will be implemented. The aid was developed using the International Patient Decision Aid Standards and is freely available. Sites randomized to this arm will require all of the HSL components as well as:
  1. Use of the Shared-Decision Aide
  2. Clinician Education on SDM
  Interventions: Other: Changes to the electronic health record (EHR); Other: Individualized audit and feedback reporting for clinicians; Other: Clinician education sessions; Other: Use of a shared decision-making (SDM) aide; Other: Shared decision-making (SDM) education

INTERVENTIONS:
Other: Changes to the electronic health record (EHR) — EHR changes will include minor changes to prescription fields to make it easier for clinicians to order "wait and see" antibiotics to be filled only if the child worsens or does not improve rather than antibiotics to take immediately.
Other: Individualized audit and feedback reporting for clinicians — Automated audit and feedback reports detailing participating clinicians' antibiotic prescribing habits for AOM both individually and in comparison to their peers will be shared with clinicians on a quarterly basis throughout the intervention period.
Other: Clinician education sessions — Virtual education sessions will be held for clinicians to learn more about national guidelines for antibiotic prescribing for AOM, etc. The sessions will be recorded and distributed to clinicians who were unable to attend. Attendance of these sessions will apply toward continuing medical education credits for participants.
Other: Use of a shared decision-making (SDM) aide — A previously validated SDM aide for AOM will be used by clinicians during visits with children with AOM. The aide will be available online and in paper form.
  Arms: Hybrid Intervention
Other: Shared decision-making (SDM) education — Clinicians will receive education on SDM and how to use the aid via virtual, recorded sessions.
  Arms: Hybrid Intervention

SUMMARY:
This study aims to improve care and reduce unnecessary antibiotic prescribing for children with ear infections. The study will compare the effectiveness of a "gold standard" to a hybrid intervention combined with this gold standard, in order to identify steps to increase parent satisfaction for child ear infection care. The "gold standard" approach is a Health System Level Intervention. On its own, it involves clinician education, tools in electronic medical records, and audit and feedback reports for clinician prescribing habits. The hybrid intervention includes the elements of the health systems level intervention in addition to a Shared Decision-Making component, which allows for both an increase in the role parents play in their child's care, as well as clinician education for how to use this method. The goals of this work are to increase parent satisfaction, reduce antibiotics taken for childhood ear infections, align medical care with the current national guidelines, and evaluate differences in the two intervention groups. Both groups will be evaluated for implementation outcomes to improve dissemination and scalability for future use of these models in antibiotic prescribing for children with ear infections.

This study will recruit a diverse group of patients and clinicians to complete surveys, parents to participate in focus groups, and clinicians and administrators to be interviewed in order to meet study aims and receive sufficient feedback on the interventions performed. There are two hypotheses for this research: 1. The Hybrid Intervention will have higher parent satisfaction and reduced antibiotic use compared to the Health-System Level Intervention and 2. The Hybrid Intervention will be more challenging to implement than the Health-System Level Intervention, but will be preferred by parents, clinicians, and administrators.

DETAILED DESCRIPTION:
Acute otitis media (AOM), commonly referred to as an ear infection, is the most common reason children are prescribed antibiotics, affecting 5 million children and resulting in 10 million antibiotic prescriptions annually. By 3 years of age over 60% of children will have had AOM. Though 84% of AOM episodes resolve without antibiotics, antibiotics are prescribed to >95% of children. The American Academy of Pediatrics (AAP) recommends that most children with AOM do not receive an immediate antibiotic (an antibiotic to take right away) and instead be managed with watchful waiting, where an antibiotic is used only if the child worsens or does not improve. In clinical trials watchful waiting reduced antibiotic use by over 62% and did not result in increased complications, reduced parent satisfaction, or increased symptoms. Unfortunately, despite these trials <5% of children with AOM are managed with watchful waiting. The use of antibiotics when not needed contributes to the development of antibiotic resistant organisms, which makes future infections more difficult to treat. Additionally, unnecessary antibiotics reduce pediatric quality of life and over 26% of children who take an antibiotic experience an adverse drug event (ADE). Thus, for every 100 children with AOM who take an antibiotic at least 26 children experience harm; whereas only 5 children have symptomatic benefit.

This study aims to compare the effectiveness of two pragmatic interventions to improve patient-centered outcomes and reduce unnecessary antibiotics taken for AOM. Interventions will be conducted at 33 community-based clinics and/or urgent care centers across three distinct geographic regions in the United States. Randomization will occur at the clinic center level to either the gold standard approach or the hybrid intervention. The Practical Robust Implementation and Sustainability Model (PRISM) will be used to guide implementation and the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework will be used to evaluate outcomes. A mixed-methods approach will be used in the pre-implementation and evaluation phases and will utilize quantitative analyses, semi-structured interviews, focus groups, and surveys.

ELIGIBILITY:
Inclusion Criteria:

A. Implementation of Interventions 1. Clinic at a participating organization 2. Provides care to children with AOM 3. Administrative or local approval for participation

B. Secondary Electronic Health Record Data

1. Aged 6 months-17-years-old (inclusive)
2. Diagnosis of AOM by ICD10 code

C. Video recordings or direct observation of the use of a shared decision aid

Parent participation:

1. Child aged 6 months-17 years (inclusive)
2. Diagnosed with AOM by clinician
3. Parent or legal guardian is present and is >=18 years or older

Clinician Participation:

1. Licensed clinician and not a medical trainee
2. Age 18 >= years or older

D. Pre-implementation interviews of clinicians and administrators

1. Licensed clinician (physician or advanced practice clinician) that cares for children with AOM at a participating organization or an administrator/manager at a participating organization.
2. Aged >=18 years-no maximum

E. Pre-implementation focus groups of parents

1. Parent or legal guardian of a child aged 6 months-17 years (inclusive) that has had AOM diagnosed at a participating organization.
2. 18 years of age or older and able/willing to consent

F. Parents enrolled for surveys

1. Parent or legal guardian of a child aged 6 months-17 years (inclusive) that has had AOM diagnosed at a participating organization. 2. Willing to participate and able to complete electronic surveys at enrollment and 10 days after enrollment. 3. Working phone 4. Age >=18 years of age

G. Post-intervention focus groups of parents

1. Parent or legal guardian of a child aged 6 months-17 years (inclusive) that has had AOM diagnosed at a participating organization.
2. 18 years of age or older and able/willing to consent

H. Post-intervention surveys of clinicians and administrators

1. Licensed clinician (physician or advanced practice clinician) that cares for children with AOM at a participating organization or an administrator/manager at a participating organization.
2. Aged >=18 years-no maximum

Exclusion Criteria:

A. Implementation of Interventions

1. Clinics that exclusively provide telehealth

B. Secondary Electronic Health Record Data

1. None

C. Video recordings or direct observation of the use of a shared decision aid

Parent participation:

1. None

Clinician Participation:

1. None

D. Pre-implementation interviews of clinicians and administrators 1. Medical trainee (student, resident, fellow, etc.)

E. Pre-implementation focus groups of parents

1. None

F. Parents enrolled for surveys 1. Complicated or recurrent AOM as determined by the study team

G. Post-intervention focus groups of parents 1. None

H. Post-intervention surveys of clinicians and administrators

1. Medical trainee (student, resident, fellow, etc.)

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1566 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Increase in Parent Satisfaction | 10 days after clinic visit for ear infection
  Survey responses will be measured by the percentage of "Very Satisfied" or "Extremely Satisfied" responses from parents on a 7-point Likert Scale. The survey tool will be created from adaptations to the Pediatric Quality of Life Inventory (PedsQL) and the Acute Otitis Media Severity of Symptom Scale (AOM-SOS). In this survey, the higher scores on the Likert Scale will indicate more overall parent satisfaction.
Percentage of Patients Taking an Antibiotic for AOM | 10 days after clinic visit for ear infection
  Comparing electronic health record prescription data with parent yes/no survey responses to a question on whether or not their child took an antibiotic prescribed for treating their ear infection.

SECONDARY OUTCOMES:
Shared Decision-Making | At time of clinic visit for ear infection (0 Days)
  Summed score of the "Knowledge and Decisional Conflict Assessment" section of the Shared Decision-Making Questionnaire (SDM Q-9). The survey has a 6-Point Likert Scale ranging in values from "Completely Disagree" to "Completely Agree". For this survey, the higher the number on the Likert Scale, the better the outcome.
Pediatric Quality of Life | 10 days after clinic visit for ear infection
  Score on the PEDS-QL Survey. This survey has a 5-Point Likert Scale ranging from "Never a Problem" (0 points) to "Almost Always a Problem" (4 points). Higher scores on this scale indicate worse outcomes while lower scores indicate better outcomes.
Symptom and Severity Duration | 0 and 10 days after clinic visit for ear infection
  Scores on a Likert scale from the AOM-Severity of Symptom scale survey on the following measures:
  1. Symptom Severity (at maximum and at 10 days)
  2. Time to Symptom Improvement (from onset)
  3. Time to All Symptom Resolution (from onset)
  4. Time to Ear Pain Resolution (from onset)
  5. Symptoms Resolved at Day 10 (yes/no)
Missed Work/School/Daycare | 10 days after clinic visit for ear infection
  Numbers of days child missed school/daycare and/or number of days parent(s) missed work
Adverse Drug Events | 10 days after clinic visit for ear infection
  Percentage of patients with adverse drug event(s)
Treatment Failure | 10 days after clinic visit for ear infection
  Percentage that changed their medication management (i.e., took an antibiotic if initially trying watchful waiting or tried a new antibiotic if initially immediately tried antibiotics)
Management Strategy | At time of clinic visit for ear infection (0 Days)
  Percentage of immediate antibiotic use
Antibiotic Prescription Filled | 10 days after clinic visit for ear infection
  Percentage of filled antibiotic prescriptions (even if not taken)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Frost, MD, Principal Investigator — Intermountain Health
Locations (3):
- United States (3):
  - Denver Health and Hospital Authority, Denver, Colorado
  - AllianceChicago, Chicago, Illinois
  - Intermountain Health, Murray, Utah

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Rinehart DJ, Gilbert A, Andersen LM, Gray TW, O'Leary S, Frost HM; DISAPEAR Study Group. Barriers and Facilitators to Implementing Watchful Waiting for Pediatric Acute Otitis Media. J Pediatr. 2025 Nov 13;289:114904. doi: 10.1016/j.jpeds.2025.114904. Online ahead of print. PMID 41241139
- [Derived] Jenkins TC, Keith A, Stein AB, Hersh AL, Narayan R, Eggleston A, Rinehart DJ, Patel PK, Walter E, Hargraves IG, Frost HM; DISAPEAR Study Group. Interventions to de-implement unnecessary antibiotic prescribing for ear infections (DISAPEAR Trial): protocol for a cluster-randomized trial. BMC Infect Dis. 2024 Jan 24;24(1):126. doi: 10.1186/s12879-023-08960-z. PMID 38267837